CLINICAL TRIAL: NCT04909086
Title: Effect of Different Modes of Isotonic Exercises on Clinical Outcomes and Cartilage Biomarkers in Knee Osteoarthritis
Brief Title: Different Modes of Isotonic Exercises for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince Sultan Military College of Health Sciences (Other)
Collaborators: King Fahd Military Medical Complex (Unknown)
Responsible Party: Principal Investigator, Ahmed Farrag, Assisstant professor, Prince Sultan Military College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAP-05-D-003
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Kinetic exercises; Biomarkers
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both the outcome assessors and the study statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Physical Therapy (Active Comparator): Control group for the study.
  Interventions: Procedure: Standard physical Therapy
- Open Kinetic Chain (Experimental): Standard care in addition to open kinetic chain exercises for the knee joint muscles.
  Interventions: Procedure: Open Kinetic Chain
- Closed Kinetic Chain (Experimental): Standard care in addition to closed kinetic chain exercises for the knee joint muscles.
  Interventions: Procedure: Closed Kinetic Chain

INTERVENTIONS:
Procedure: Standard physical Therapy — Patients assigned to this group will receive a 40-min multimodal supervised physical therapy treatment comprised of warm-up (10-min cycling/walking), muscle stretching, neuromuscular control exercises, and ten-minute transcutaneous electrical nerve stimulation (TENS). Manual mobilization techniques may be applied as necessary according to the findings of the physical examination. Treating physical therapists will prescribe exercises based on a predetermined list of exercises.
  Arms: Standard Physical Therapy
Procedure: Closed Kinetic Chain — Patients assigned to this group will receive a 40-min multimodal supervised physical therapy treatment comprised of warm-up (10-min cycling/walking), three sets of 10 repetitions of 60% of one-repetition maximum (1RM) of seated leg press and partial squat exercises, neuromuscular control exercises, and ten-minute transcutaneous electrical nerve stimulation (TENS). Manual mobilization techniques may be applied as necessary according to the findings of the physical examination. Treating physical therapists will prescribe exercises based on a predetermined list of exercises.
  Arms: Closed Kinetic Chain
Procedure: Open Kinetic Chain — Patients assigned to this group will receive a 40-min multimodal supervised physical therapy treatment comprised of warm-up (10-min cycling/walking), three sets of 10 repetitions of 60% of one-repetition maximum (1RM) of Quadriceps seated strengthening and Hamstring curl-up exercises, neuromuscular control exercises, and ten-minute transcutaneous electrical nerve stimulation (TENS). Manual mobilization techniques may be applied as necessary according to the findings of the physical examination. Treating physical therapists will prescribe exercises based on a predetermined list of exercises.
  Arms: Open Kinetic Chain

SUMMARY:
This is a randomized controlled trial examining and compare the effects of open and closed kinetic chain exercises on pain, function, and cartilage synthesis and degradation biomarkers after an eight-week rehabilitation program for knee osteoarthritis (OA) patients.

DETAILED DESCRIPTION:
Design and Subjects: A prospective, active control, three-parallel-group, assessor-blinded, randomized controlled trial. A sample of 120 subjects will be recruited and randomly assigned to one of three study groups at a 1:1:1 allocation ratio (40 participants per group): a) Standard care only, b) Closed kinetic chain exercises plus standard care, and c) Open kinetic chain plus standard care.

Intervention: participants will receive 24 treatment sessions (3 sessions/week) over 8 weeks. Participants will be allocated to the experimental groups will receive the standard care protocol in addition to either closed or open-chain exercises.

Outcome measures: The primary outcomes are physical function and pain assessed using the Western Ontario and McMaster Universities (WOMAC) scores. Secondary outcomes include the Numeric Pain Rating Scale, quadriceps and hamstring strength, joint range of motion (ROM), joint proprioception error, and serum and urine OA biomarkers including the Serum cartilage oligomeric matrix protein (COMP), Serum propeptide Type-II N-terminal (PIIANP), Serum C- reactive protein (CRP), and Urine type -II Collagen telopeptide (CTX-II).

Data Analysis: Data will be analyzed using the intension-to-treat (ITT) analysis with multiple imputations. The primary analysis of the primary outcomes at a two-month follow-up time point (after completing the intervention protocol for 8 weeks) will be carried out using a mixed-model analysis of variance (ANOVA) test with adjustment for a set of pre-specified baseline factors. Secondary analysis using the ANOVA test for the primary outcomes at a six-month follow-up time point, and secondary outcomes at all follow-up time points will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years of age;
* having knee pain;
* having at least three of the following additional symptoms: a-morning stiffness ≤ 30 minutes, b-crepitation, c-bone margin tenderness, d-bony enlargement or e-no palpable warmth;
* willing to provide informed consent

Exclusion Criteria:

* Knee joints showing Kellgren and Lawrence (K-L) grades 1 or 4;
* rheumatoid arthritis;
* serious pathological conditions (inflammatory arthritis and malignancy); total or partial arthroplasty of the affected knee joint, or on a waiting list for joint replacement surgery;
* recent surgical procedure of the lower extremities in the previous 6 months;
* uncontrolled hypertension and unstable cardiovascular problems that could subject the participant to increased risk with exercise and physical exertion;
* physical incapability to safely perform exercises, walking or stationary cycling, as in debilitating visual defects, neurological problems, exaggerated low back pain, advanced osteoporosis, and inability to walk 10 meters without an assistive device;
* use of prescribed analgesics, corticosteroid or analgesic injection intervention for knee pain within the previous 30 days;
* lack of clear comprehension of study procedures or inability to comply with instructions;
* stated inability to attend or complete the proposed course of intervention and follow-up schedule.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain score using the Arabic version of the Western Ontario and McMaster Universities (WOMAC) index | Baseline, 2, and 6 months follow-up
  A 5-point Likert scale comprised of 24 questions across 3 subscales. Standardized answers are assigned a score from 0 (no symptoms) to 4 (extreme symptoms) with higher scores indicating worst pain, stiffness, and function.
Change in function score using the Arabic version of the Western Ontario and McMaster Universities (WOMAC) index | Baseline, 2, and 6 months follow-up
  A 5-point Likert scale comprised of 24 questions across 3 subscales. Standardized answers are assigned a score from 0 (no symptoms) to 4 (extreme symptoms) with higher scores indicating worst pain, stiffness, and function.

SECONDARY OUTCOMES:
Change in knee pain using the Arabic version of the Numeric Pain Rating Scale (ANPRS) | Baseline, 2, and 6 months follow-up
  A horizontal 11-point scale (0-10), with 0 indicating no pain and 10 indicating the worst pain ever.
Change in isometric muscle strength | Baseline, 2, and 6 months follow-up
  Measured in Newtons for the Quadriceps and Hamstring muscles using a hand-held dynamometer (Commander Muscle testing, JTech, USA). The greater the recorded value the better the muscle strength.
Change in knee joint range of motion (ROM) | Baseline, 2, and 6 months follow-up
  Active knee joint flexion/extension ROM measured in degrees using an electric goniometer (Biometrics Ltd, DLK900, UK). The greater the recorded value the greater the knee joint ROM.
Change in knee joint proprioception | Baseline, 2, and 6 months follow-up
  Active repositioning error of a given passive position of the knee joint will be assessed using an electric goniometer (Biometrics Ltd, DLK900, UK). The lesser the recorded value the better the knee joint proprioception.
Change in knee OA biomarkers | Baseline, 2, and 6 months follow-up
  Serum (10 ml blood) and urine samples will be collected from the participants and analyzed using the Enzyme-linked immunosorbent assay (ELISA) technique.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Farrag, PhD, Principal Investigator — Prince Sultan Military College of Health Sciences
Locations (1):
- King Fahd Military Medical Complex, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No